CLINICAL TRIAL: NCT04378387
Title: Usefulness of the Ipsilateral and Contralateral Index for the Interpretation of Adrenal Vein Sampling (AVS) in the Subtype Diagnosis of Primary Aldosteronism
Brief Title: Ipsilateral and Contralateral Index for the Interpretation of Adrenal Vein Sampling (AVS) in Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Mauro Maccario, Medical Doctor, Professor, University of Turin, Italy
Other Study IDs: ICI-AVS
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral)
Keywords: Primary Aldosteronism; Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism Due to Adrenal Hyperplasia (Bilateral); Adrenal Vein Sampling; Renin-Angiotensin-Aldosterone System; Blood Pressure; Lateralization Index; Ipsilateral Index; Contralateral Index
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adrenal vein sampling (AVS) is currently considered the gold standard for subtype diagnosis of primary aldosteronism (PA). However, the percentage of unsuitable procedures due to the unsuccessful cannulation of one of the two adrenal veins is still considerable, and there is no general consensus on the criteria that should be used for the interpretation of the results of an AVS study in these specific cases.

DETAILED DESCRIPTION:
The differentiation between subtypes of primary aldosteronism (PA) is fundamental to refer each patient to the most appropriate therapeutic approach (surgical in case of unilateral disease and medical in case of bilateral disease). Adrenal vein sampling (AVS) is currently considered the gold standard for such differentiation between subtypes.

However, despite significant progress in optimizing the AVS procedure, the percentage of unsuitable procedures due to the unsuccessful cannulation of one of the two adrenal veins is still considerable, especially in less experienced centers.

It would therefore be important to identify criteria for the interpretation of the results of a suboptimal AVS study (i.e. with sampling of only one of the two adrenal veins). This problem has recently been addressed by some groups; however, there is still no general consensus on these criteria and all existing studies must be considered exploratory in this field.

In this study, therefore, all patients with PA followed by our center and who underwent a successful (i.e. with correct cannulation and sampling from both adrenal veins) unstimulated (i.e. without cosyntropin stimulation) AVS procedure will be retrospectively evaluated.

If a reliable unilateral index could be identified for subtype diagnosis, this tool could be used for the interpretation of suboptimal AVS data, thus preventing a certain percentage of patients from the necessity to repeat the procedure and allowing to refer each one, also on the basis of an incomplete dataset, to the most appropriate therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Diagnosis of Primary Aldosteronism
* Execution of Adrenal Vein Sampling (AVS) for Subtype Diagnosis

Exclusion Criteria:

* Execution of AVS in stimulated condition (i.e. with cosyntropin stimulation)
* Inability to achieve successful catheterization of one or both adrenal veins during AVS (as established by adrenal/peripheral vein cortisol ratio)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients followed by our center with age over 18 years old and a diagnosis of primary aldosteronism, who underwent a successful (i.e. with successful catheterization of both adrenal veins) unstimulated adrenal vein sampling between January 2005 and April 2020.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Monolateral index for each adrenal gland in each patient | At AVS procedure
  For each adrenal gland, monolateral index will be computed by dividing the ratio of aldosterone/cortisol in its adrenal vein by the ratio of aldosterone/cortisol in a peripheral vein. By definition, this will be a unitless index. The index will be compared between three main groups of interest (i.e. adrenal glands with a final diagnosis of ipsilateral Conn adenoma, adrenal glands with a final diagnosis of contralateral Conn adenoma, adrenal glands with a final diagnosis of bilateral adrenal hyperplasia).
Aldosterone/cortisol index for each adrenal gland in each patient | At AVS procedure
  For each adrenal gland, aldosterone/cortisol index represents the ratio of aldosterone/cortisol in its adrenal vein. Aldosterone will be measured in pg/ml, cortisol will be measured in mcg/l. The index will be compared between three main groups of interest (i.e. adrenal glands with a final diagnosis of ipsilateral Conn adenoma, adrenal glands with a final diagnosis of contralateral Conn adenoma, adrenal glands with a final diagnosis of bilateral adrenal hyperplasia).

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Maccario, MD, Principal Investigator — Endocrinology, Diabetology and Metabolism; University of Turin; Ezio Ghigo, MD, Study Chair — Endocrinology, Diabetology and Metabolism; University of Turin
Locations (1):
- Division of Endocrinology, Diabetology and Metabolism; University of Turin, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Background] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Background] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Background] Pasternak JD, Epelboym I, Seiser N, Wingo M, Herman M, Cowan V, Gosnell JE, Shen WT, Kerlan RK Jr, Lee JA, Duh QY, Suh I. Diagnostic utility of data from adrenal venous sampling for primary aldosteronism despite failed cannulation of the right adrenal vein. Surgery. 2016 Jan;159(1):267-73. doi: 10.1016/j.surg.2015.06.048. Epub 2015 Oct 2. PMID 26435431
- [Background] Fujii Y, Umakoshi H, Wada N, Ichijo T, Kamemura K, Matsuda Y, Kai T, Fukuoka T, Sakamoto R, Ogo A, Suzuki T, Nanba K, Tsuiki M, Naruse M; WAVES-J Study Group. Subtype prediction of primary aldosteronism by combining aldosterone concentrations in the left adrenal vein and inferior vena cava: a multicenter collaborative study on adrenal venous sampling. J Hum Hypertens. 2017 Dec;32(1):12-19. doi: 10.1038/s41371-017-0015-0. Epub 2017 Nov 24. PMID 29176594
- [Background] Lee BC, Chang CC; TAIPAI Study Group. Regarding "Diagnostic utility of data from adrenal venous sampling for primary aldosteronism despite failed cannulation of the right adrenal vein". Surgery. 2016 May;159(5):1478-9. doi: 10.1016/j.surg.2015.10.033. Epub 2015 Dec 17. No abstract available. PMID 26706611
- [Background] Strajina V, Al-Hilli Z, Andrews JC, Bancos I, Thompson GB, Farley DR, Lyden ML, Dy BM, Young WF, McKenzie TJ. Primary aldosteronism: making sense of partial data sets from failed adrenal venous sampling-suppression of adrenal aldosterone production can be used in clinical decision making. Surgery. 2018 Apr;163(4):801-806. doi: 10.1016/j.surg.2017.10.012. Epub 2017 Nov 22. PMID 29174432
- [Background] Wang TS, Kline G, Yen TW, Yin Z, Liu Y, Rilling W, So B, Findling JW, Evans DB, Pasieka JL. A Multi-institutional Comparison of Adrenal Venous Sampling in Patients with Primary Aldosteronism: Caution Advised if Successful Bilateral Adrenal Vein Sampling is Not Achieved. World J Surg. 2018 Feb;42(2):466-472. doi: 10.1007/s00268-017-4327-6. PMID 29124355